CLINICAL TRIAL: NCT03127423
Title: Comparison Between One-stage Hybrid Ablation and Thoracoscopic Surgical Ablation for Intractable Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-828
Record Dates: First submitted 2016-12-03; First posted 2017-04-25 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Hybrid ablation; Thoracoscope
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Hybrid ablation group (Experimental): Patients in this group will receive one-stop intervention with totally thoracoscopic surgical ablation and percutaneous catheter ablation.
  Interventions: Procedure: Hybrid ablation
- Thoracoscopic surgical ablation group (Active Comparator): Patients in this group will receive only totally thoracoscopic surgical ablation with Fuwai lesion set.
  Interventions: Procedure: Thoracoscopic surgical ablation

INTERVENTIONS:
Procedure: Hybrid ablation — This intervention includes totally thoracoscopic surgical ablation and percutaneous catheter ablation simultaneously.
  Arms: Hybrid ablation group
Procedure: Thoracoscopic surgical ablation — This intervention only includes totally thoracoscopic surgical ablation without percutaneous catheter ablation.
  Arms: Thoracoscopic surgical ablation group

SUMMARY:
Previous evidence indicated that the outcomes of both video-assisted thoracoscopic surgical ablation and percutaneous radiofrequency ablation therapy for persistent atrial fibrillation (AF) were unsatisfied. Recently, hybrid ablation therapy for AF had encouraging outcomes. However, there were no randomized, controlled clinical studies to prove the effectiveness of this new strategy. This study is aimed to compare the outcomes of hybrid ablation with video-assisted thoracoscopic surgical ablation for persistent AF with enlarged left atrium.

DETAILED DESCRIPTION:
This study is aimed to compare the outcomes of hybrid ablation with video-assisted thoracoscopic surgical ablation for persistent AF with enlarged left atrium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one anti-arrhythmic drugs
* Persistent AF lasting more than 1 year or with a left atrial diameter>50mm

Exclusion Criteria:

* Previous percutaneous catheter ablation or surgical ablation
* Presence of significant structural heart disease (dilated cardiomyopathy, hypertrophic cardiomyopathy, valvular heart disease, untreated coronary artery disease)
* Left atrial diameter>60mm
* Previous thoracic or lung operation
* Left atrial thrombosis or left atrial appendage thrombosis
* Chronic obstructive pulmonary disease (COPD) (Forced expiratory volume in 1 second (FEV1)/Forced vital capacity (FVC)<70%、FEV1<50% anticipated value)
* Bilateral carotid artery stenosis>80%
* Refuse to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Survival rate without any recurrence of AF | At 12-month after intervention
  Without detections of AF (episodes longer than 30 seconds)

SECONDARY OUTCOMES:
Burden of AF | At 12-month after intervention
  Burden of AF according to Tele-ECG-Card lasting for one week
Quality of life score | preoperative and 12-month after intervention
  Measured with questionnaire of AF effect on Quality of Life
Adverse events | 12 months follow up
  Major adverse cardiovascular events; Major bleeding events; Major thromboembolic events.
Left atrial function | preoperative and postoperative
  left atrial ejection fraction and left atrial expansion index
postoperative complications | 30 days after operation
  perioperative complication of catheter ablation and thoracoscopic surgical abaltion
Survival rate without any recurrence of atrial tachyarrhythmia | At 12-month after intervention
  Survival rate without AF, atrial flutter or atrial tachycardia will be defined by absence of any of these electrocardiographically documented events lasting > 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD,PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No